CLINICAL TRIAL: NCT06862310
Title: Effect of Lactobacillus- and Bifidobacterium-containing Yogurt on Gut Microbiota and Short-chained Fatty Acids
Brief Title: Effects of Fermented Dairy Products on Defecation Changes Through Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Z-Plus Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: lin5611_1; A-109-082 (Other: Taipei Medical University)
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Defecation Irregularity
Keywords: defecation; yogurt; Lactobacillus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): acidified milk without adding beneficial bacteria
  Interventions: Other: yogurt intervention
- yogurt intervention (Experimental): probiotic-enriched fermented milk (2.0 × 10⁹ Colony-forming unit [CFU]/mL)
  Interventions: Other: yogurt intervention

INTERVENTIONS:
Other: yogurt intervention — daily probiotics dose of 3 × 108 CFU (95% confidence interval [CI]: 1 × 109 to 3 × 1010 CFU) in 112 mL of fermented milk per day (95% CI: 100-187.5 mL/day)

SUMMARY:
The investigators recruited participants aged 20-65 years who did not have gastrointestinal diseases and who were not taking medication for digestive symptoms (e.g., gastric acid inhibitors, antibiotics, sterilization medications, or antidiarrheal agents) in the month before enrollment. The participants were prohibited from consuming any probiotic foods, supplements, or fermented dairy products except those that were provided during the 6-week study. Each participant first completed a 2-week adaptation period (n = 22). Subsequently, each participant was randomly assigned to either a control or intervention group. The participants received two 200-g daily servings of either a probiotic-infused fermented milk or a control dairy product for 4 weeks.

DETAILED DESCRIPTION:
This single-center, double-blind, parallel-design clinical trial assessed the impact of a probiotics-containing fermented milk consumed daily for 4 weeks on defecation patterns and the composition of the gut microbiome in healthy adults. We recruited participants aged 20-65 years who did not have gastrointestinal diseases and who were not taking medication for digestive symptoms (e.g., gastric acid inhibitors, antibiotics, sterilization medications, or antidiarrheal agents) in the month before enrollment. The participants were prohibited from consuming any probiotic foods, supplements, or fermented dairy products except those that were provided during the 6-week study. Each participant first completed a 2-week adaptation period (n = 22). Subsequently, each participant was randomly assigned to either a control or intervention group. The participants received two 200-g daily servings of either a probiotic-infused fermented milk or a control dairy product for 4 weeks. The intervention product contained 2 × 109 colony-forming units (CFU)/mL of Lactobacillus acidophilus and Bifidobacterium lactis, along with two starter cultures of Streptococcus thermophilus and L. bulgaricus. The intervention group was administered a median daily probiotics dose of 3 × 108 CFU (95% confidence interval [CI]: 1 × 109 to 3 × 1010 CFU) in 112 mL of fermented milk per day (95% CI: 100-187.5 mL/day). A written consent was obtained from each participant prior to the initiation of this study. The randomized controlled trial protocol was approved by the Joint Institutional Review Board of Taipei Medical University, Taiwan (N202101006 and N202110014).

Baseline Characteristics and Food Records Anthropometric and blood measurement data were collected at baseline and after 4 weeks of intervention. These included body weight, height, body mass index, lipid profile, and levels of liver function markers. Three-day food records (two weekdays and one weekend day) were collected at baseline and during each of the 4 weeks of intervention to monitor the participants' dietary habits.

Defecation frequency and constipation symptoms Since the selected subjects were healthy individuals, defecation frequency per week and Bristol Stool Scale scores were assessed using a questionnaire given to the participants.

Fecal Microbiota Analysis Fecal samples were collected at baseline and after the intervention. We used selective media, prepared as described elsewhere, to analyze the concentrations of Bifidobacterium spp., Lactobacillus spp., C. perfringens, and coliform organisms in the fecal samples. Five participants were randomly selected from each group, and their microbiome compositions were analyzed using 16S rRNA sequencing. Briefly, bacterial genomic DNA was isolated from the participants' stool samples using the QIAamp Fast DNA Stool Mini Kit (QIAGEN, Germany), and the V3-V4 region of bacterial 16S rRNA genes was amplified using universal primers (341F and 805R). Demultiplexed paired reads were processed using Cutadapt software, v1.12 (DOI:10.14806/ej.17.1.200), and the filtered reads were analyzed using the DADA2 package, v1.3.5, in R software, v3.3.3, following the workflow proposed by Callahan et al. but without rarefying.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-65 years old
* without gastrointestinal diseases or other health problems
* agree not to consume antibiotics, health supplements that may affect the composition of intestinal flora (ex. probiotics, prebiotics), and fermented dairy products (ex. yogurt, cheese other than those provided in this experiment) during the experiment.

Exclusion Criteria:

* under pregnancy
* with gastrointestinal diseases or other health problems

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Defecation frequency per week | From enrollment to the end of treatment at 4 weeks
  defecation frequency per week was recorded by the participients

SECONDARY OUTCOMES:
Participant feeling during defecation | From enrollment to the end of treatment at 4 weeks
  verbal (written) description of the feeling of straining, feel of stool texture, and feeling of constipation

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
results not been published yet